CLINICAL TRIAL: NCT05007106
Title: A Multicenter, Open-label, Phase 2 Basket Study of MK-7684A, a Co-formation of Vibostolimab (MK-7684) With Pembrolizumab (MK-3475), With or Without Other Anticancer Therapies in Participants With Selected Solid Tumors
Brief Title: MK-7684A With or Without Other Anticancer Therapies in Participants With Selected Solid Tumors (MK-7684A-005) (KEYVIBE-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7684A-005; MK-7684A-005 (Other: MSD); jRCT2031210335 (Registry Identifier: jRCT); KEYVIBE-005 (Other: MSD); 2023-505284-36-00 (Registry Identifier: EU CT); U1111-1291-4290 (Registry Identifier: UTN); 2021-001009-56 (EudraCT Number)
Record Dates: First submitted 2021-08-10; First posted 2021-08-16 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Uterine Cervical Neoplasms; Endometrial Neoplasms; Squamous Cell Carcinoma of Head and Neck; Gallbladder Neoplasms; Cholangiocarcinoma; Esophageal Neoplasms; Triple Negative Breast Neoplasms; Hepatocellular Carcinoma; Urinary Bladder Neoplasms; Ovarian Neoplasms; Stomach Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Squamous Cell Carcinoma of Head and Neck; Gallbladder Neoplasms; Cholangiocarcinoma; Esophageal Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Hepatocellular; Urinary Bladder Neoplasms; Ovarian Neoplasms; Stomach Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib; Fluorouracil; Cisplatin; Paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Carboplatin; Docetaxel; Bevacizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Participants with locally recurrent unresectable or metastatic cervical cancer whose tumors express programmed cell death 1 ligand 1 (PD-LI) and have a combined positive score (CPS) ≥1 will be randomly assigned to treatment with either pembrolizumab/vibostolimab co-formulation or pembrolizumab only. The other study intervention arms will be assigned to participants depending on the selected cancer type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Pembrolizumab/Vibostolimab Co-Formulation (Experimental): Participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous (IV) infusion every 3 weeks (Q3W) up to 35 cycles. Participants receiving pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) will be given the option to transition to pembrolizumab monotherapy.
  Interventions: Biological: Pembrolizumab/Vibostolimab Co-Formulation; Biological: Pembrolizumab
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg via IV infusion Q3W up to 35 cycles.
  Interventions: Biological: Pembrolizumab
- Pembrolizumab/Vibostolimab Co-Formulation + Lenvatinib (Endometrial Cancer Cohort) (Experimental): Participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion Q3W up to 35 cycles, plus lenvatinib 20 mg once daily (qd) up to 45 cycles. Participants receiving pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) will be given the option to transition to pembrolizumab monotherapy in combination with Lenvatinib.
  Interventions: Biological: Pembrolizumab/Vibostolimab Co-Formulation; Biological: Pembrolizumab; Drug: Lenvatinib
- Pembrolizumab/Vibostolimab Co-Formulation + Lenvatinib (Hepatocellular Cancer Cohort) (Experimental): Participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via intravenous IV infusion Q3W up to 35 cycles, plus lenvatinib 12 mg (body weight [BW] ≥60 kg) or lenvatinib 8 mg (BW <60 kg) qd up to 45 cycles. Participants receiving pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) will be given the option to transition to pembrolizumab monotherapy in combination with Lenvatinib.
  Interventions: Biological: Pembrolizumab/Vibostolimab Co-Formulation; Biological: Pembrolizumab; Drug: Lenvatinib
- Pembrolizumab/Vibostolimab + 5-Fluorouracil + Cisplatin (Experimental): Participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via IV infusion Q3W, plus 5-fluorouracil (5-FU), plus Cisplatin as background therapy. Participants receiving pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) will be given the option to transition to pembrolizumab monotherapy in combination with 5-Fluorouracil + Cisplatin.
  Interventions: Biological: Pembrolizumab/Vibostolimab Co-Formulation; Biological: Pembrolizumab; Drug: 5-Fluorouracil; Drug: Cisplatin
- Pembrolizumab/Vibostolimab Co-Formulation + Paclitaxel (Experimental): Participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via IV infusion Q3W up to 35 cycles, plus paclitaxel as background therapy until meeting discontinuation criteria. Participants receiving pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) will be given the option to transition to pembrolizumab monotherapy in combination with Paclitaxel.
  Interventions: Biological: Pembrolizumab/Vibostolimab Co-Formulation; Biological: Pembrolizumab; Drug: Paclitaxel
- Pembrolizumab/Vibostolimab Co-Formulation + Gemcitabine/Cisplatin (Experimental): Participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via IV infusion Q3W up to 35 cycles, plus gemcitabine (until disease progression or unacceptable toxicity) and cisplatin (up to 8 cycles) as background therapy. Participants receiving pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) will be given the option to transition to pembrolizumab monotherapy in combination with Gemcitabine/Cisplatin
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: Gemcitabine
- Pembrolizumab/Vibostolimab Co-Formulation+ Carboplatin/Paclitaxel/Bevacizumab (Experimental): Participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via IV infusion Q3W up to 35 cycles, plus carboplatin, paclitaxel, and bevacizumab as local standard of care (SOC) background therapy. Participants receiving pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) will be given the option to transition to pembrolizumab monotherapy in combination with Carboplatin/Paclitaxel/Bevacizumab.
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin; Drug: Docetaxel; Drug: Bevacizumab
- Pembrolizumab/Vibostolimab Co-Formulation + Capecitabine/Oxaliplatin (Experimental): Participants receive pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) via IV infusion Q3W up to 35 cycles, plus capecitabine and oxaliplatin as background therapy. Participants receiving pembrolizumab/vibostolimab (coformulation of 200 mg pembrolizumab and 200 mg vibostolimab) will be given the option to transition to pembrolizumab monotherapy in combination with Capecitabine/Oxaliplatin.
  Interventions: Biological: Pembrolizumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Biological: Pembrolizumab/Vibostolimab Co-Formulation — Pembrolizumab 200 mg plus vibostolimab 200 mg administered via IV infusion Q3W
  Other Names: MK-7684A
  Arms: Pembrolizumab/Vibostolimab + 5-Fluorouracil + Cisplatin; Pembrolizumab/Vibostolimab Co-Formulation; Pembrolizumab/Vibostolimab Co-Formulation + Lenvatinib (Endometrial Cancer Cohort); Pembrolizumab/Vibostolimab Co-Formulation + Lenvatinib (Hepatocellular Cancer Cohort); Pembrolizumab/Vibostolimab Co-Formulation + Paclitaxel
Biological: Pembrolizumab — Pembrolizumab 200 mg administered via IV infusion Q3W.
  Other Names: MK-3475; KEYTRUDA®
Drug: Lenvatinib — Lenvatinib 20 mg, 12 mg, or 8 mg (dependent on cancer type and body weight) administered via oral capsule QD
  Other Names: Lenvima; E7080; MK-7902
  Arms: Pembrolizumab/Vibostolimab Co-Formulation + Lenvatinib (Endometrial Cancer Cohort); Pembrolizumab/Vibostolimab Co-Formulation + Lenvatinib (Hepatocellular Cancer Cohort)
Drug: 5-Fluorouracil — 5-FU 800 mg/m^2/day administered via continuous IV infusion on each of days 1 to 5 Q3W for up to 35 cycles
  Other Names: 5-FU; Fluracil
  Arms: Pembrolizumab/Vibostolimab + 5-Fluorouracil + Cisplatin
Drug: Cisplatin — Cisplatin administered via IV infusion
  Other Names: Platinol; cis Platinum
  Arms: Pembrolizumab/Vibostolimab + 5-Fluorouracil + Cisplatin; Pembrolizumab/Vibostolimab Co-Formulation + Gemcitabine/Cisplatin
Drug: Paclitaxel — Paclitaxel administered via IV infusion at investigator's choice of dose
  Other Names: Taxol; Abraxane; Anzatax
  Arms: Pembrolizumab/Vibostolimab Co-Formulation + Paclitaxel; Pembrolizumab/Vibostolimab Co-Formulation+ Carboplatin/Paclitaxel/Bevacizumab
Drug: Gemcitabine — Gemcitabine administered via IV infusion on Day 1 and Day 8 of each 3-week cycle, until PD or unacceptable toxicity
  Arms: Pembrolizumab/Vibostolimab Co-Formulation + Gemcitabine/Cisplatin
Drug: Carboplatin — Carboplatin administered via IV infusion at investigator's choice of dose and frequency
  Arms: Pembrolizumab/Vibostolimab Co-Formulation+ Carboplatin/Paclitaxel/Bevacizumab
Drug: Docetaxel — For participants who cannot receive paclitaxel due to hypersensitivity or adverse event (AE), docetaxel administered via IV infusion Q3W, Day 1 of each cycle for up to 5 cycles
  Arms: Pembrolizumab/Vibostolimab Co-Formulation+ Carboplatin/Paclitaxel/Bevacizumab
Drug: Bevacizumab — Bevacizumab (or biosimilars such as MVASI®, Zirabev®, Aybintio®, ALYMSYS®, Abevmy®, Onbevezy®, Vegzelma®) administered via IV infusion Q3W; Day 1 of each 3-week cycle for up to 15 cycles
  Arms: Pembrolizumab/Vibostolimab Co-Formulation+ Carboplatin/Paclitaxel/Bevacizumab
Drug: Capecitabine — Capecitabine administered via oral tablet twice daily on Days 1 to 14 of each cycle (Q3W) for up to 35 cycles
  Arms: Pembrolizumab/Vibostolimab Co-Formulation + Capecitabine/Oxaliplatin
Drug: Oxaliplatin — Oxaliplatin administered via IV infusion Q3W up to 35 cycles
  Arms: Pembrolizumab/Vibostolimab Co-Formulation + Capecitabine/Oxaliplatin

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and preliminary efficacy of pembrolizumab/vibostolimab co-formulation (MK-7684A) with or without other anticancer therapies in participants with selected advanced solid tumors. The primary hypothesis is that pembrolizumab/vibostolimab co-formulation is superior to pembrolizumab alone in terms of objective response rate or progression-free survival in participants with cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* One of the following histologically or cytologically confirmed, advanced (unresectable or metastatic) solid tumors:

  * Squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix
  * Endometrial cancer
  * Head and neck squamous cell carcinoma (HNSCC)
  * Unresectable biliary adenocarcinoma (gallbladder or biliary tree [intrahepatic or extrahepatic] cholangiocarcinoma)
  * Adenocarcinoma or squamous cell carcinoma of the esophagus or advanced/metastatic Siewert type 1 adenocarcinoma of the gastroesophageal junction (GEJ).
  * Triple-negative breast cancer (TNBC)
  * Hepatocellular carcinoma (HCC)
  * Urothelial carcinoma of the renal pelvis, ureter, bladder, or urethra
  * Ovarian cancer
  * Gastric cancer
* Measurable disease per RECIST v1.1 as assessed by BICR or local site investigator.
* Adequately controlled blood pressure (BP) with or without antihypertensive medications.
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on anti-retroviral therapy (ART).
* Male participants must agree to follow contraceptive guidance.
* Female participants are not pregnant or breastfeeding, not a woman of child-bearing potential (WOCBP) or is a WOCBP and agrees to follow contraceptive guidance.
* Adequate organ function.

Exclusion Criteria:

* History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 3 years.
* Prior therapy with anti-programmed cell-death (PD-1), anti-PD-L1, anti-PD-L2, or anti-T-cell immunoreceptor with Ig and ITIM domains (TIGIT) agent.
* Prior systemic anticancer therapy including investigational agents within 4 weeks before randomization/allocation.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of study medication.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* Active infection requiring systemic therapy.
* Concurrent active hepatitis B and hepatitis C virus infection.
* History of allogenic tissue/solid organ transplant.
* Previous treatment with lenvatinib (for participants who will receive lenvatinib in their assigned treatment arm).
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 2 years
  ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience a CR or PR as assessed by blinded independent central review based on RECIST 1.1 will be presented.
Progression-Free Survival (PFS) per RECIST 1.1 as Assessed by BICR | Up to approximately 2 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
ORR per RECIST 1.1 as Assessed by Investigator in Participants with Selected Solid Tumors | Up to approximately 2 years
  ORR is defined as the percentage of participants who have a CR (Disappearance of all target lesions) or a PR (At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience a CR or PR as assessed by investigator based on RECIST 1.1 will be presented.
PFS per RECIST 1.1 as Assessed by Investigator at 9 months | 9 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.
PFS per RECIST 1.1 as Assessed by Investigator at 12 months | 12 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 5.5 years
  OS is defined as the time from randomization to death due to any cause.
PFS per RECIST 1.1 as Assessed by Investigator | Up to approximately 2 years
  PFS is defined as the time from first dose of study treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by investigator will be presented.
Duration of Response (DOR) per RECIST 1.1 as Assessed by BICR | Up to approximately 2 years
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or confirmed PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The DOR as assessed by BICR will be presented.
DOR per RECIST 1.1 as Assessed by Investigator | Up to approximately 2 years
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or confirmed PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The DOR as assessed by investigator will be presented.
ORR per RECIST 1.1 as Assessed by Investigator | Up to approximately 2 years
  ORR is defined as the percentage of participants who have a CR (Disappearance of all target lesions) or a PR (At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience a CR or PR as assessed by investigator based on RECIST 1.1 will be presented.
PFS per RECIST 1.1 as Assessed by Investigator in Participants with Cervical Cancer | Up to approximately 2 years
  PFS is defined as the time from first dose of study treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by investigator will be presented.
Change from Baseline in Global Health Status/Quality of Life Score (European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 [EORTC QLQ-C30] Items 29 and 30) | Baseline and up to approximately 2 years
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined score will be presented.
Change from Baseline in Physical Functioning Score (EORTC QLQ-C30 Items 1-5) | Baseline and up to approximately 2 years
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better quality of life. The change from baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) score will be presented.
Number of Participants Who Experienced One or More Adverse Events (AEs) | Up to approximately 2 years
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Number of Participants Who Discontinued Study Intervention Due to an AE | Up to approximately 2 years
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (73):
- United States (14):
  - Alaska Womens Cancer Care ( Site 1016), Anchorage, Alaska
  - City of Hope Comprehensive Cancer Center ( Site 1001), Duarte, California
  - University of California, Irvine (UCI) Health - UC Irvine Me-Chao Family Comprehensive Cancer Cente, Orange, California
  - Karmanos Cancer Institute ( Site 1007), Detroit, Michigan
  - Memorial Sloan Kettering - Basking Ridge ( Site 1023), Basking Ridge, New Jersey
  - Memorial Sloan Kettering - Monmouth ( Site 1022), Middletown, New Jersey
  - Memorial Sloan Kettering - Bergen ( Site 1025), Montvale, New Jersey
  - Memorial Sloan Kettering- Commack ( Site 1021), Commack, New York
  - Memorial Sloan Kettering - Westchester ( Site 1020), Harrison, New York
  - Memorial Sloan Kettering Cancer Center ( Site 1002), New York, New York
  - Memorial Sloan Kettering - Nassau ( Site 1026), Uniondale, New York
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 1024), Tulsa, Oklahoma
  - Sanford Cancer Center-Gynecologic Oncology ( Site 1015), Sioux Falls, South Dakota
  - Houston Methodist Hospital ( Site 1017), Houston, Texas
- Canada (2):
  - Kingston Health Sciences Centre-Kingston General Hospital Site ( Site 1051), Kingston, Ontario
  - Princess Margaret Cancer Centre ( Site 1056), Toronto, Ontario
- Chile (4):
  - FALP-UIDO ( Site 1401), Santiago, Region M. de Santiago
  - Oncovida ( Site 1405), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 1402), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 1404), Temuco, Región de la Araucanía
- Colombia (5):
  - Fundacion Colombiana de Cancerología Clinica Vida ( Site 1422), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 1421), Barranquilla, Atlántico
  - Instituto Nacional de Cancerología-Clinical Oncology ( Site 1425), Bogotá, Cundinamarca
  - Oncologos del Occidente ( Site 1424), Pereira, Risaralda Department
  - Fundación Cardiovascular de Colombia ( Site 1423), Piedecuesta, Santander Department
- France (6):
  - CENTRE LEON BERARD-Medical oncology ( Site 1151), Lyon, Auvergne-Rhône-Alpes
  - Centre Georges François Leclerc ( Site 1155), Dijon, Cote-d Or
  - Institut Regional du Cancer Montpellier ( Site 1157), Montpellier, Herault
  - Gustave Roussy-medicine departement ( Site 1153), Villejuif, Paris
  - Sainte Catherine Institut du Cancer Avignon Provence-Oncologie médicale ( Site 1156), Avignon, Vaucluse
  - Institut Curie ( Site 1152), Paris
- Germany (5):
  - Universitaetsklinikum Heidelberg-Nationales Centrum für Tumorerkrankungen ( Site 1180), Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen-Department of Internal Medicine VIII - Medical Oncology, ECTU, Pne, Tübingen, Baden-Wurttemberg
  - Klinikum der Universität München Großhadern ( Site 1176), München, Bavaria
  - Universitaetsklinikum Duesseldorf-Gastroenterology, Hepatology and Infectiology ( Site 1172), Düsseldorf, North Rhine-Westphalia
  - Charite Universitätsmedizin Berlin Campus Benjamin Franklin ( Site 1171), Berlin
- Israel (4):
  - Rambam Health Care Campus-Oncology ( Site 1141), Haifa
  - Hadassah Medical Center-Oncology ( Site 1142), Jerusalem
  - Sheba Medical Center-ONCOLOGY ( Site 1144), Ramat Gan
  - Sourasky Medical Center-Oncology ( Site 1143), Tel Aviv
- Italy (5):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Ginecologia Oncologica ( Site 1136), Rome, Lazio
  - Ospedale San Raffaele-Oncologia Medica ( Site 1135), Milan, Lombardy
  - Istituto Clinico Humanitas-U.O di Oncologia medica ed Ematologia ( Site 1138), Rozzano, Milano
  - Istituto Europeo di Oncologia IRCCS-Divisione di Sviluppo di Nuovi Farmaci per Terapie Innovative (, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-S.C. Sperimentazioni Cliniche ( Site 1134), Napoli
- Japan (4):
  - Aichi Cancer Center Hospital ( Site 1324), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 1321), Kashiwa, Chiba
  - Osaka International Cancer Institute ( Site 1323), Osaka
  - National Cancer Center Hospital ( Site 1322), Tokyo
- Netherlands (2):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek - NKI-AVL ( Site 1121), Amsterdam, North Holland
  - Erasmus Medisch Centrum-Medical Oncology ( Site 1122), Rotterdam, South Holland
- Poland (3):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Oddzial Badan Wczesnych Faz ( Site 1101, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 1103), Gdansk, Pomeranian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 1104), Koszalin, West Pomeranian Voivodeship
- South Korea (3):
  - Seoul National University Hospital-Internal Medicine ( Site 1312), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 1311), Seoul
  - Asan Medical Center ( Site 1313), Seoul
- Spain (5):
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals-Medical Oncology ( Site 1113), Hospitalet, Barcelona
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 1117), Pozuelo de Alarcón, Madrid
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 1111), Madrid, Madrid, Comunidad de
  - Clinica Universidad de Navarra-Medical Oncology ( Site 1118), Madrid
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO ( Site 1114), Seville
- Taiwan (4):
  - NATIONAL CHENG-KUNG UNI. HOSP.-clinical trial center ( Site 1302), Tainan
  - National Taiwan University Hospital-Oncology ( Site 1301), Taipei
  - Mackay Memorial Hospital ( Site 1305), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 1304), Taoyuan District
- Turkey (Türkiye) (7):
  - Istanbul Universitesi Cerrahpasa ( Site 1203), Istanbul- Fatih, Istanbul
  - Baskent University Dr. Turgut Noyan Research and Training Center ( Site 1201), Adana
  - Hacettepe Universitesi-oncology hospital ( Site 1209), Ankara
  - Ankara City Hospital-Medical Oncology ( Site 1202), Ankara
  - Trakya University-Medical Oncology ( Site 1207), Edirne
  - Acibadem Universitesi Atakent Hastanesi ( Site 1208), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1204), Istanbul

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26136&tenant=MT_MSD_9011